CLINICAL TRIAL: NCT00167843
Title: A Longitudinal Study Assessing the Infectious Status and Immunity of Mothers and Their Children in Lambaréné, Including Intermittent Treatment of Children With Sulfadoxine-pyrimethamine for Malaria Control and Its Impact on Long-term Health
Brief Title: Reducing the Effects of Malaria in Children by Administering Repeated Preventive Doses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Albert Schweitzer Hospital (Other)
Collaborators: Medical Research Unit, Lambarene (Unknown); Bundesministerium fuer Bildung und Forschung (BMBF) (Unknown); Deutscher Akademischer Austausch Dienst (Other); German Research Foundation (Other); Bill and Melinda Gates Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 28574
Record Dates: First submitted 2005-09-11; First posted 2005-09-14 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Malaria
Keywords: Malaria; Anemia; Children; Gabon; Intermittent preventive treatment
MeSH Terms: conditions — Malaria; Anemia | interventions — fanasil, pyrimethamine drug combination

INTERVENTIONS:
Drug: sulfadoxine-pyrimethamine

SUMMARY:
The general goal of the project is to assess the infectious status and immunity of mothers and children living in a malaria region. A major part of the study involves administering an effective antimalarial, sulfadoxine-pyrimethamine (Fansidar®), to children at the same timepoints as vaccinations, i.e. at age 3, 9 and 15 months. The main objective is to study safety, efficacy, and consequences of such a strategy in particular the ability to reduce the risk of anemia.

DETAILED DESCRIPTION:
More than 1.5 million deaths of African children under 5 years of age are due to Plasmodium falciparum malaria. There is an urgent need for available and affordable strategies to control malaria morbidity in childhood.

Malaria control measures have been assessed for their potential to reduce intensity of infection in order to decrease the risk of malaria. It has been shown that malaria prevention using drugs is potentially capable to reduce malaria morbidity, school absenteeism, and all-cause mortality. However, prevention using drugs in the first years of life can also result in the loss or delay of acquired resistance which can lead to a rebound phenomenon (i.e. an increased risk of severe malaria after the therapy ended). In a recent study on intermittent treatment with Fansidar® at 2, 3, and 9 months of age, the number of malaria cases during the first 12 months of life was significantly reduced and no rebound effect was observed. This study has demonstrated that the intermittent administration of Fansidar® is safe and has beneficial effects for the children. However, the effectiveness decreased some months after discontinuing the drug. The promising effect of the intermittent administration of fansidar shown in this study needs to be confirmed in areas of different endemicity such as Lambaréné, Gabon. It is assumed that a more extended intermittent application of Fansidar® than performed in the above example would likely result in a longer period of protection from malaria, and the extended intermittent administration of Fansidar should not lead to rebound effects resulting in a higher occurrence of malaria.

The framework of this study offers a unique opportunity to study characteristics of infectious disease of importance in the Lambaréné area and the development of resistance against microbes at the maternofetal (mother/foetus) interface. Comparable studies will simultaneously take place in two associated study sites (Kumasi and Tamale) with different malaria endemicity in Ghana, West Africa.

Comparison: Comparison of malaria attacks in children with and without intermittent Fansidar® treatment with drug administration at months 3 and 9 (alongside with routine vaccinations delivered through child vaccination programme) and an additional administration at month 15.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Permanent residence in the study area

Exclusion Criteria:

* Allergy/hypersensitivity to sulfonamides or pyrimethamine
* Signs of severe hepatic or renal dysfunction not due to malaria

Max Age: 5 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1189
Dates: Start 2002-12; Study Completion 2007-03

PRIMARY OUTCOMES:
Efficacy:
The proportion of children with at least one episode of anemia from 3 to 18 months of life
The proportion of children with at least one episode of malaria from 3 to 18 months of life
Safety:
The proportion of children with at least one episode of an adverse event
The proportion of children with at least one episode of a serious adverse event
Rebound:
The proportion of children with at least one episode of anemia from 18-30 months of life, the proportion of children with at least one episode of malaria from 18-30 months of life

SECONDARY OUTCOMES:
Proportion of children with at least one episode of severe anemia
Proportion of hospitalized children with anemia
Proportion of hospitalized children with malaria
Proportion of hospitalized children with any disease
Proportion of children with at least one episode of anemia from 3 to 12 months of life
Proportion of children with at least one episode of malaria from 3 to 12 months of life.
Parasite drug resistance after intermittent sulfadoxine-pyrimethamine and placebo application
Multiplicity of P. falciparum infections after the intermittent treatment
Antibody responses against variable parasite genes after the intermittent treatment
Specific responses to malaria vaccine candidates during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Peter G Kremsner, MD, Principal Investigator — Albert Schweitzer Hospital
Locations (1):
- Medical Research Unit of the Albert Schweitzer Hospital, Lambaréné, Moyen-Ogooué Province, Gabon

REFERENCES:
- [Background] WHO. In WHO report: Fostering Development, Geneva, 1996
- [Background] Greenwood BM, Greenwood AM, Bradley AK, Snow RW, Byass P, Hayes RJ, N'Jie AB. Comparison of two strategies for control of malaria within a primary health care programme in the Gambia. Lancet. 1988 May 21;1(8595):1121-7. doi: 10.1016/s0140-6736(88)91949-6. PMID 2896957
- [Background] Menendez C, Kahigwa E, Hirt R, Vounatsou P, Aponte JJ, Font F, Acosta CJ, Schellenberg DM, Galindo CM, Kimario J, Urassa H, Brabin B, Smith TA, Kitua AY, Tanner M, Alonso PL. Randomised placebo-controlled trial of iron supplementation and malaria chemoprophylaxis for prevention of severe anaemia and malaria in Tanzanian infants. Lancet. 1997 Sep 20;350(9081):844-50. doi: 10.1016/S0140-6736(97)04229-3. PMID 9310602
- [Background] Schellenberg D, Menendez C, Kahigwa E, Aponte J, Vidal J, Tanner M, Mshinda H, Alonso P. Intermittent treatment for malaria and anaemia control at time of routine vaccinations in Tanzanian infants: a randomised, placebo-controlled trial. Lancet. 2001 May 12;357(9267):1471-7. doi: 10.1016/S0140-6736(00)04643-2. PMID 11377597
- [Background] Bradley-Moore AM, Greenwood BM, Bradley AK, Bartlett A, Bidwell DE, Voller A, Kirkwood BR, Gilles HM. Malaria chemoprophylaxis with chloroquine in young Nigerian children. I. Its effect on mortality, morbidity and the prevalence of malaria. Ann Trop Med Parasitol. 1985 Dec;79(6):549-62. doi: 10.1080/00034983.1985.11811962. PMID 3914860
- [Background] Diagne N, Rogier C, Sokhna CS, Tall A, Fontenille D, Roussilhon C, Spiegel A, Trape JF. Increased susceptibility to malaria during the early postpartum period. N Engl J Med. 2000 Aug 31;343(9):598-603. doi: 10.1056/NEJM200008313430901. PMID 10965006
- [Derived] Gabor JJ, Schwarz NG, Esen M, Kremsner PG, Grobusch MP. Dengue and chikungunya seroprevalence in Gabonese infants prior to major outbreaks in 2007 and 2010: A sero-epidemiological study. Travel Med Infect Dis. 2016 Jan-Feb;14(1):26-31. doi: 10.1016/j.tmaid.2016.01.005. Epub 2016 Jan 29. PMID 26869532
- [Derived] Grobusch MP, Gabor JJ, Aponte JJ, Schwarz NG, Poetschke M, Doernemann J, Schuster K, Koester KB, Profanter K, Borchert LB, Kurth F, Pongratz P, Issifou S, Lell B, Kremsner PG. No rebound of morbidity following intermittent preventive sulfadoxine-pyrimethamine treatment of malaria in infants in Gabon. J Infect Dis. 2009 Dec 1;200(11):1658-61. doi: 10.1086/647990. PMID 19848610
- [Derived] May J, Adjei S, Busch W, Gabor JJ, Issifou S, Kobbe R, Kreuels B, Lell B, Schwarz NG, Adjei O, Kremsner PG, Grobusch MP. Therapeutic and prophylactic effect of intermittent preventive anti-malarial treatment in infants (IPTi) from Ghana and Gabon. Malar J. 2008 Oct 1;7:198. doi: 10.1186/1475-2875-7-198. PMID 18828899
- [Derived] Grobusch MP, Lell B, Schwarz NG, Gabor J, Dornemann J, Potschke M, Oyakhirome S, Kiessling GC, Necek M, Langin MU, Klein Klouwenberg P, Klopfer A, Naumann B, Altun H, Agnandji ST, Goesch J, Decker M, Salazar CL, Supan C, Kombila DU, Borchert L, Koster KB, Pongratz P, Adegnika AA, Glasenapp Iv, Issifou S, Kremsner PG. Intermittent preventive treatment against malaria in infants in Gabon--a randomized, double-blind, placebo-controlled trial. J Infect Dis. 2007 Dec 1;196(11):1595-602. doi: 10.1086/522160. Epub 2007 Oct 25. PMID 18008242
- See also: Homepage of IPTi consortium — http://www.ipti-malaria.org
- See also: Homepage of the Medical Research Unit of the Albert Schweitzer Hospital — http://www.lambarene.org